CLINICAL TRIAL: NCT03934827
Title: A First in Human, Phase 1 Safety Study in Two Parts to Determine the Safety, Tolerability and Anti-cancer Immune-modulatory Effects of MRx0518 in Patients With Solid Tumour Awaiting Surgical Removal of the Tumour.
Brief Title: MRx0518 in Patients With Solid Tumours Waiting Surgical Removal of the Tumour
Acronym: MICROBIOME
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Collaborators: 4D pharma plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: C/35/2017
Record Dates: First submitted 2019-04-15; First posted 2019-05-02 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Melanoma; Breast Cancer; Uterine Cancer; Ovarian Cancer; Prostate Cancer; Urethral Cancer; Bladder Cancer; Renal Cancer; Lung Cancer; Head and Neck Cancer
Keywords: Cancer; Solid Tumour
MeSH Terms: conditions — Melanoma; Breast Neoplasms; Uterine Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Urethral Neoplasms; Urinary Bladder Neoplasms; Kidney Neoplasms; Lung Neoplasms; Head and Neck Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: 20 participants will receive open label MRx0518 in an initial preliminary safety phase. A further 100 participant will then receive MRx0518/Placebo in a 4:1 ratio in a double blinded randomised phase.
Who Masked: Participant, Investigator
Masking Description: Part A: open Label; Part B: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Open label, preliminary phase
  20 participants
  Interventions: Drug: MRx0518 Capsules
- Part B (Experimental): Randomised, double blinded phase
  100 participants
  Interventions: Drug: MRx0518/placebo Capsules

INTERVENTIONS:
Drug: MRx0518 Capsules — MRx0518 is a live biotherapeutic product consisting of a lyophilised formulation of a proprietary strain of bacterium. The dosing regimen is one capsule orally twice daily for 2-4 weeks until surgery.
  Arms: Part A
Drug: MRx0518/placebo Capsules — MRx0518/placebo product consist of a lyophilised formulation of either a proprietary strain of bacterium or placebo.The dosing regimen is one capsule orally twice daily for 2-4 weeks until surgery. Placebo capsules are manufactured to mimic MRx0518 capsules and contain the same excipients as the active biotherapeutic product.
  Arms: Part B

SUMMARY:
The primary objective is to determine the safety and tolerability of the novel compound, MRx0518 in patients with solid tumours at 30 days post-surgery.

20 participants will receive open label MRx0518 in a preliminary safety phase. After successful evaluation by the Independent Safety Monitoring Committee (IDMC), a further 100 participants will be recruited to receive MRx0518/Placebo.

DETAILED DESCRIPTION:
This is a first in human, single centre study in two parts, which aims to determine the safety and tolerability of the novel biotherapeutic compound, MRx0518, to examine its use as an anti-cancer and immune system modulating agent in patients with a range of solid tumours, over 2 years.

MRx0518 is composed of a proprietary strain of bacterium (Enterococcus species) which is found in the gastrointestinal tract of approx. 25% of humans and is predicted, from preclinical studies, to produce beneficial effects in humans.

Patients who have been diagnosed with melanoma, breast, ovarian, uterine, prostate, urethra, bladder, renal, lung or head and neck cancer, who are amenable to surgical resection, will receive MRx0518 (part A) or MRx0518/placebo (part B) orally twice daily for 2-4 weeks until surgery to remove the tumour. In part A, 20 patients will receive open label MRx0518 as part of a preliminary safety assessment. Following surgery, patients will attend a 30 day, 6 month, 12 month and 24 month follow up visit.

Following successful evaluation of part A data by the Independent Data Monitoring Committee (IDMC) the study will continue to recruit a further 100 patients to Part B of the trial. Part B will be placebo controlled, in which patients will be randomised in a double blinded fashion in a 4:1 ratio of MRx0518:placebo. In total, 120 patients will be recruited into the study (20 from part A and 100 from part B).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or over
2. Provide written (signed and dated) informed consent and be capable of understanding the study and co-operating with treatment and follow-up.
3. Have radiologically, histologically or cytologically confirmed melanoma, breast, ovarian, uterine, prostate, urethra, bladder, renal, lung, or head and neck cancer* that is considered amenable to primary surgical resection and where primary surgery is planned but would not routinely have been performed until 2-4 weeks post initial biopsy.*New primary cancers or recurrences are permissible provided the patient has not received chemotherapy, radiotherapy or surgery for the last two years prior to screening.
4. Have a life expectancy of greater than 12 weeks.
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status 0-2
6. Have normal organ and marrow function.
7. Women of child-bearing potential and men must agree to use adequate and highly effective contraception for at least 28 days prior to dosing until one complete menstrual cycle post dosing for women and 3 months after the last dose for men. Alternatively, true abstinence may be used, where this is in line with the preferred and usual lifestyle of the patient.
8. Able to swallow and retain oral medication.

Exclusion Criteria:

1. Patients who have had any anti-cancer therapy within the last 2 years.
2. Patients with cancer affecting the gastrointestinal tract or those where bowel resection is considered to be highly likely to be required.
3. Patients may not be receiving any other investigational agents or receiving concurrent anti-cancer therapy. In addition, all herbal (alternative) medicines are excluded.
4. Patients not willing, or for whom it is not planned, to undergo primary surgery for their cancer 2-4 weeks after initiation of therapy with IMP.
5. Patient who would otherwise have undergone primary surgery within 2 weeks of starting therapy with IMP.
6. Patients who have rapidly progressive local disease, or local disease that, in the opinion of the investigator, is not amenable to surgical resection.
7. Patients with known structural or valvular heart valve defects, gastrointestinal fistula, feeding tubes and inflammatory bowel disease or those who are immunosuppressed or receiving immunosuppressant medication (steroids up to an equivalent dose of 20mg of prednisolone daily is allowed as long as the dose has been stable for the last 6 months).
8. Patients who smoke or use nicotine in any form including e-cigarettes and nicotine patches or sprays or have smoked/used nicotine in the 3 months prior to screening.
9. Patients who consume more than 14 units of alcohol per week, on a regular basis.
10. History of allergic reactions attributed to compounds of similar biologic composition to MRx0518.
11. Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, including patients with active hepatitis B virus (HBV), active hepatitis C virus (HCV) who have a detectable viral load, and patients with Human Immunodeficiency Virus (HIV), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations, gastrointestinal disease that would limit compliance with study requirements.
12. Any significant infection e.g. influenza, fever over 38°C, meningitis or an infection resulting in the subject seeking a consultation with a healthcare professional, within four weeks of starting IMP therapy.
13. Pregnant women are excluded from this study because teratogenic or abortifacient effects are unknown. Furthermore, there is an unknown but potential risk for adverse events in nursing infants, secondary to treatment of the mother with MRx0518 so breastfeeding should be discontinued if the mother is treated with MRx0518.
14. Patients with gastrointestinal disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis).
15. Patients who have completed a course of antibiotics within the four weeks before dosing.
16. Patients who are allergic to amoxicillin/clavulanic acid, erythromycin and imipenem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of MRx0518 as determined through the collection of the number and severity of adverse vents (AEs) and serious adverse events (SAEs). | Baseline upto 30 days post surgery.
  AEs and SAEs will be assessed by CTCAE v5.0
Safety and tolerability of MRx0518 determined by clinically significant changes in biochemistry, haematology and urinalysis laboratory results. | Baseline upto 30 days post surgery.
  Assessed by clinically significant changes in biochemistry results (albumin, bilirubin, urea, creatinine, total protein, c reactive protein, calcium, chloride, sodium, phosphorus, potassium, bicarbonate, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, gamma-glutamyl-transferase, globulin, lactate dehydrogenase, creatine kinase, cholesterol, triglycerides, uric acid, and fasting glucose); haematology results (haemoglobin, platelets, RBC, haematocrit, WBC, neutrophils, lymphocytes, monocytes, eosinophils, basophils) and urinalysis results (occult blood, glucose, protein, ketones, nitrite, leucocytes, pH and specific gravity).
Safety and tolerability of MRx0518 determined by clinically significant changes in vital signs. | Baseline upto 30 days post surgery.
  Assessed by the measurement of pulse, blood pressure, temperature and respiratory rate.
Safety and tolerability of MRx0518 as determined by clinically significant changes in electrocardiogram (ECG) results. | Baseline upto 30 days years post surgery.
  Assessed by the measurement of RR interval, PR interval, QRS duration, QT interval and QTc interval.
Safety and tolerability of MRx0518 as determined by clinically significant changes upon physical examination. | Baseline upto 30 days post surgery.
  Assessed by clinically significant abnormal changes to the general appearance, skin, head and neck, lymph nodes, thyroid, musculoskeletal/extremities, cardiovascular, respiratory, abdomen and neurological assessment.

SECONDARY OUTCOMES:
Response of MRx0518 determined by the measurement of tumour markers. | Baseline (optional) and during surgery.
  Tissue biopsies taken at screening (optional) and during surgery and analysed for tumour biomarkers (e.g. Ca125 in gynaecological malignancies, Ca153 in breast cancer).
Overall survival of patients who receive MRx0518 compared to placebo. | Survival of subjects will be recorded up to 2 years post-surgery
  Survival of individual patients will be assessed from the start of treatment until death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Jonathan Krell, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No